CLINICAL TRIAL: NCT06861738
Title: Comaring the Effect of Paracetamol in Tratment of Headach
Brief Title: Effect of Parcetamol in Headach
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Bazied Dardir mohamed, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: parasetamol in headach
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Headache
Keywords: paracetamol
MeSH Terms: conditions — Headache | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): patients will recive paracetamol
  Interventions: Drug: Paracetamol (acetaminophen)
- groupB (Placebo Comparator): patients will recive placebo
  Interventions: Drug: Paracetamol Placebo

INTERVENTIONS:
Drug: Paracetamol (acetaminophen) — oral paracetamol 500mg three times per day
  Arms: Group A
Drug: Paracetamol Placebo — placebo tab three time per day
  Arms: groupB

SUMMARY:
Tension-type headache (TTH) affects about 1 person in 5 worldwide. It is divided into infrequent episodic TTH (fewer than one headache per month), frequent episodic TTH (two to 14 headaches per month), and chronic TTH (15 headache days a month or more). Paracetamol (acetaminophen) is one of a number of analgesics suggested for acute treatment of headaches in frequent episodic TTH.Objectives To assess the efficacy and safety of paracetamol for the acute treatment of frequent episodic TTH in adults.

DETAILED DESCRIPTION:
Headaches are a commonly reported problem in community-based surveys worldwide. The lifetime prevalence of headache is estimated to be greater than 90% , and the annual prevalence rate is estimated to be 46% in the general adult population . Variations in reported prevalence may result from differences in study design, population, inclusion or exclusion of cases of infrequent episodic TTH, overlap with probable migraine, cultural and environmental differences, or even genetic factors . TTH is more common than migraine, a finding replicated across the work.

The management of people with headaches is largely neglected , and may be fragmented by the involvement of clinicians from different medical specialities (neurology; ear, nose and throat; ophthalmology; psychiatry). Because headache is rarely life-threatening and headache pain is generally mild to moderate in intensity, people often self medicate and do not seek formal care from health services .

Headache can be either primary (no underlying cause) or secondary (due to other systemic or local causes) . TTH belongs to the group of primary headaches and is seen in nearly one-third of people experiencing headaches; the large number of people affected imposes a significant burden on the healthcare system. Generally, episodes of TTH are mild to moderate in intensity, and self limiting, but in a small group of people they may be more severe and disabling . People with longer lasting or more severe headaches may seek help in a clinical setting, but the majority of people do not do so, resulting often in inadequate and inappropriate management .

ELIGIBILITY:
Inclusion Criteria:

* both sex
* 18 years old to 65 years
* free ct brain

Exclusion Criteria:

* migrane
* any brain pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
pain score VAS score | 24 hours
  VAS Score for pain

IPD SHARING:
Plan to Share IPD: Undecided